CLINICAL TRIAL: NCT04729673
Title: Canine Occlusal Relationship Changes After Full Mouth Rehabilitation and Stainless-Steel Crown Placement Under General Anesthesia in A Group of Egyptian Children; Part 2: "A Before and After Study"
Brief Title: Canine Occlusal Relationship Changes After Full Mouth Rehabilitation Under General Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Nourhan Kamal, Principal Investigator, Cairo University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 14422019435625
Record Dates: First submitted 2021-01-25; First posted 2021-01-28 (Actual); Last update posted 2023-08-09 (Actual); Status verified 2023-08

CONDITIONS: General Anesthesia
Keywords: Full mouth rehabilitation; Canine Overlap relation; vertical dimension of occlusion; canine occlusal relation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patient's normal canine occlusal relationship. (Active Comparator): Before full mouth rehabilitation with stainless steel crowns for primary molars , the vertical dimension of occlusion from gingival zenith of upper and lower primary canines shall be determined at the right and left sides. The distance shall be determined using a digital caliper.(Shenzhen Jiabaili Electronic Commerce Co., Ltd), and the reading will be photographed by a digital camera (iPhone 11 dual 12 MP Ultra-Wide and wide camera,Apple Inc.).
  Interventions: Device: Digital caliper (Shenzhen Jiabaili Electronic Commerce Co., Ltd)
- Canine occlusal relation after full mouth rehabilitation (Sham Comparator): After full mouth rehabilitation with stainless steel crowns for primary molars , the vertical dimension of occlusion from gingival zenith of upper and lower primary canines shall be determined at the right and left sides. The distance shall be determined using a digital caliper.(Shenzhen Jiabaili Electronic Commerce Co., Ltd), and the reading will be photographed by a digital camera (iPhone 11 dual 12 MP Ultra-Wide and wide camera,Apple Inc.).
  Interventions: Device: Digital caliper (Shenzhen Jiabaili Electronic Commerce Co., Ltd)

INTERVENTIONS:
Device: Digital caliper (Shenzhen Jiabaili Electronic Commerce Co., Ltd) — Measuring the vertical distance between the gingival zenith of the upper canine to the gingival zenith of the lower canine

SUMMARY:
The aim of the study is to assess and compare canine occlusal relation in children with carious primary molars before they are treated by stainless steel crowns under general anesthesia and after their placement ,to evaluate the possibility and the time required for the post operative canine relation to resolve and how the treatment affects frequency and type of food intake.

DETAILED DESCRIPTION:
1. Children who require immediate full mouth rehabilitation under general anaesthesia will be recruited from the General Anesthesia (GA) unit in the Department of Pediatric Dentistry, Faculty of Oral and Dental Medicine, Cairo University.
2. Two postgraduate students will be filling the patient's assessment chart as shown in appendices prior to treatment. They will measure the canine occlusal relation. The measurements will be made in the maximum intercuspation position (MIP) in the centric occlusion (CO) guided by the operators' hand.
3. Before general anesthesia, an anesthesiologist and an internal medicine specialist will examine participating children, and the necessary preclinical tests will be requested.
4. On the day of the procedure, parents of the participants will fill a questionnaire asking for previous dental treatments of the child and his/her medical history and acceptance to join the study (written consent).
5. The canine occlusal relationship of both upper and lower primary canines shall be determined by measuring the vertical dimension from the gingival zenith of the upper canine and the gingival zenith of the lower canine at the right and left sides.
6. The distance shall be determined using a digital caliper (Shenzhen Jiabaili Electronic Commerce Co., Ltd), and the reading will be photographed by a digital camera (iPhone 11 dual 12 MP Ultra-Wide and wide camera, Apple Inc.).
7. For further accuracy, this will be repeated twice, and in case of the presence of a difference, the measurement will be repeated for the third time, and the mean of the values will be calculated.
8. The treatment will be performed under general anesthesia, tooth preparation will be done, and the eight Stainless-steel Crowns (3M™ ESPE™ Stainless Steel Primary Molar Crowns) will be seated.
9. The measured values will be recorded preoperatively and immediately after the treatment while the patient is unconscious.
10. Pre-operative determination of the canine occlusal relation of the upper and lower primary canines will be done; after placement during the operation and after 1, 2 and 6 months follow up period.

ELIGIBILITY:
Inclusion Criteria:

* Medical history: normal healthy children with no physical or mental disorders.
* Gender: No sex predilection.
* Age: children from (2 to 6) years old showing uncooperative behavior.
* Teeth: Carious teeth requiring oral dental rehabilitation under general requiring SSCs placement for primary molars.

Exclusion Criteria:

* Children with special health care needs or with systemic conditions
* Decayed primary canines with severe caries involving more than one-third of the incisal and palatal surfaces, class IV or V, crowns being built up or any incisal edge involvement.
* Parafunctional occlusion, i.e., Crossbite.
* Erupted permanent first molar.
* Malocclusion.
* Refusal of participation.

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 73 (Actual)
Dates: Start 2021-07-03 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
Change in the canine occlusal relationship | Day 1
  The change of the canine occlusal relationship in millimeters using digital caliper

SECONDARY OUTCOMES:
The time needed for the bite to re-adapt | ''1 month"
  The time needed for the bite to re-adapt throughout days using digital caliper
The time needed for the bite to re-adapt | ''2 months"
  The time needed for the bite to re-adapt throughout days using digital caliper
The time needed for the bite to re-adapt | ''6 months"
  The time needed for the bite to re-adapt throughout days using digital caliper

CONTACTS AND LOCATIONS:
Overall Officials: PhD, Study Director — Cairo University
Locations (1):
- Cairo University, Giza, Select A State Or Province, Egypt

IPD SHARING:
Plan to Share IPD: No